CLINICAL TRIAL: NCT06192290
Title: Home-based Transitional Telerehabilitation in Cardiac Recovery: A Study on the Health-Related Quality of Life and Therapeutic Self-Care in Older Adults Post Coronary Artery Bypass Grafting
Brief Title: Home-based Transitional Telerehabilitation in Cardiac Recovery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Hashem El-Monshed, Associate Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Home-based TT in Cardiac Rec.
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Cardiac Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): (1) aged 60 years or older; (2) diagnosed with CAD and were recommended to undergo elective CABG by a cardiologist; (3) intact cognitive function; (4) agree to be visited by the researchers at home; and (5) didn't have previous experiences with CABG. These Patients receive the usual care only.
- Intervention Group (Experimental): (1) aged 60 years or older; (2) diagnosed with CAD and were recommended to undergo elective CABG by a cardiologist; (3) intact cognitive function; (4) agree to be visited by the researchers at home; and (5) didn't have previous experiences with CABG. These Patients will receive the Video film presentations and content (16 parts)
  Interventions: Behavioral: Home-based transitional Cardiac Telerehabilitation

INTERVENTIONS:
Behavioral: Home-based transitional Cardiac Telerehabilitation — This comprehensive series is divided into 16 parts, each addressing crucial aspects of open-heart surgery recovery. Part 1 introduces open-heart surgery, heart disease symptoms, and preoperative preparations for elderly patients. Part 2 delves into cardiac rehabilitation, defining objectives and detailing recovery stages. Part 3 covers care for surgical incisions and infection signs. Part 4 explores sleep and rest, while Part 5 guides patients on a healthy post-surgery diet. Part 6 focuses on nursing interventions for dyspnea, and Part 7 addresses post-surgery cough. Part 8 discusses nursing interventions for thrombosis prevention
  Arms: Intervention Group

SUMMARY:
The main aim is to determine the impact of home video-based cardiac rehabilitation program on elderly patients' health-related quality of life and therapeutic self-care post-coronary revascularization

DETAILED DESCRIPTION:
Over the past decade, the efficacy of coronary artery bypass graft (CABG) surgery in treating coronary artery disease (CAD) has significantly advanced, particularly in improving symptom relief and survival rates among older adults. Remarkably, CAD stands as the foremost cause of global mortality, contributing to a staggering 16% of all deaths, with a notable surge of more than 2 million additional fatalities recorded in 2019, reaching a total of 8.9 million. This escalating incidence is particularly pronounced in the Middle East and North Africa, where CAD has witnessed a 160% increase, signifying a critical healthcare concern with a mortality rate of 120 per 100,000 individuals.

In the realm of cardiovascular diseases, individuals aged 75 years and above face substantial threats, with CAD posing a significant threat to both morbidity and mortality. Despite the acknowledged benefits of CABG, older adults' post-CABG commonly grapple with a spectrum of musculoskeletal and neurological challenges stemming from the surgical procedure. This encompasses incisional sternotomy pain, respiratory issues, weakness, leg swelling, sleeping difficulties, wound healing complications, poor appetite, dissatisfaction with postoperative supportive care, and difficulties with eating. Psycho-socially, these individuals often experience distress, depression, a sense of loss of control, concerns about surgery success, social dysfunction, and fear of death.

The postoperative period necessitates an in-hospital stay of approximately one week, with depressed functional capacity immediately following CABG, potentially linked to fear of activity and pain exacerbated by movement. This is followed by a convalescence period of 2 to 6 weeks for recovery after discharge and the resumption of daily activities. The healing process for chest and leg wounds typically spans 4 to 6 weeks, with pulmonary function and lung capacity decreasing one week following CABG up to 4-6 months after surgery compared to pre-surgery levels.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older
* diagnosed with CAD and were recommended to undergo elective CABG by a cardiologist
* intact cognitive function
* agree to be visited by the researchers at home
* didn't have previous experiences with CABG.

Exclusion Criteria:

* Have an experience with CABG
* demonstrates cognitive dysfunctions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Coronary revascularization outcome questionnaire (CROQ)- CROQ-CABG version | through study completion, an average of 1 year
  Developed by schroter S and Lamping DL (2004) (34) to be the only practical and scientifically validated patient-based measure of outcome for coronary revascularization that is acceptable to patients, the only tool that includes psychosocial and cognitive functioning as well as surgery-specific items, and satisfies rigorous psychometric criteria for reliability, validity, and responsiveness. This validated instrument developed specifically for use before and after CABG and PTCA, which is quick and easy to administer and provides more appropriate content as it contains items directly addressing the impact of these procedures based on problems that patients reported to be important.

SECONDARY OUTCOMES:
The Sidani Doran Therapeutic Self-Care Measure (SDTSCM) -The Home Setting care Version | through study completion, an average of 1 year
  Developed by Sidani and Doran (2001) & (2002) (35,36). to measure the action taken by a patient to promote, maintain or improve health, prevent sickness, detect and manage symptoms, and regain normal functioning. This 12-item scale measures a person's ability to perform activities that are directed at maintaining health, managing health, and restoring function (37). Patients were asked to rate their ability to perform self-care activities when home (38), with a 6-point numeric rating scale anchored with "not at all (0)" and "very much (5)".

CONTACTS AND LOCATIONS:
Locations (1):
- Shark El-Madinah Hospital, the Secretariat of Specialized Medical Centers (Cardiothoracic Surgery Department and Intensive Care Unit), Alexandria, Egypt

REFERENCES:
- [Result] Ghisi GL, Grace SL, Thomas S, Oh P. Behavior determinants among cardiac rehabilitation patients receiving educational interventions: an application of the health action process approach. Patient Educ Couns. 2015 May;98(5):612-21. doi: 10.1016/j.pec.2015.01.006. Epub 2015 Jan 20. PMID 25638305
- [Result] Fosbol EL, Zhao Y, Shahian DM, Grover FL, Edwards FH, Peterson ED. Repeat coronary revascularization after coronary artery bypass surgery in older adults: the Society of Thoracic Surgeons' national experience, 1991-2007. Circulation. 2013 Apr 23;127(16):1656-63. doi: 10.1161/CIRCULATIONAHA.113.001882. Epub 2013 Mar 26. PMID 23532630
- [Result] Osailan A, Abdelbasset WK. Exercise-based cardiac rehabilitation for postcoronary artery bypass grafting and its effect on hemodynamic responses and functional capacity evaluated using the Incremental Shuttle Walking Test: A retrospective pilot analysis. J Saudi Heart Assoc. 2020 Apr 17;32(1):25-33. doi: 10.37616/2212-5043.1005. eCollection 2020. PMID 33154888
- [Result] Lim SK, Han JY, Choe YR. Comparison of the Effects of Cardiac Rehabilitation Between Obese and Non-obese Patients After Acute Myocardial Infarction. Ann Rehabil Med. 2016 Oct;40(5):924-932. doi: 10.5535/arm.2016.40.5.924. Epub 2016 Oct 31. PMID 27847723